CLINICAL TRIAL: NCT04449991
Title: Per-protocol Repeat Kidney Biopsy in Incident Cases of Lupus Nephritis
Acronym: REBIOLUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Ioannis Parodis, Principle Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REBIOLUP
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Lupus Nephritis
Keywords: systemic lupus erythematosus; lupus nephritis; kidney biopsy; renal function impairment; long-term prognosis; electron microscopy
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: At baseline, patients will be randomised 1:1 to either undergo or not undergo a per-protocol repeat kidney biopsy at month 12 from baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm: Repeat kidney biopsy at M12 (Experimental): Patients will undergo repeat kidney biopsy at month 12 from baseline.
  Interventions: Procedure: Repeat kidney biopsy
- Control arm: No repeat kidney biopsy (No Intervention): Patients will not undergo repeat kidney biopsy at month 12 from baseline.

INTERVENTIONS:
Procedure: Repeat kidney biopsy — Intensification of immunosuppression if NIH AI > 3
  Arms: Intervention arm: Repeat kidney biopsy at M12

SUMMARY:
Lupus nephritis (LN) is one of the most severe complications of systemic lupus erythematosus (SLE). Among people living with SLE, 35-60% will develop LN during the course of the disease. This complication is one of the factors that contribute to deterioration of the renal function.

Some centres perform kidney biopsies after completion of treatment for an episode of LN as a part of the treatment evaluation. The term "repeat biopsy" is often used to describe these biopsies. Several studies have reported that repeat kidney biopsies show activity at the level of tissue, even in patients with normal routine blood and urine markers. The investigators strongly believe that this information is important, and should be taken into consideration during decision of treatment. To provide evidence for this, the investigators have designed a collaborative project within the frame of the Lupus Nephritis Trials Network. With this research project, the investigators want to contribute to an increased proportion of patients with LN who achieve remission (inactivity) of LN, and a reduced proportion of patients who worsen in renal function in the long term.

Patients with SLE who develop a first episode of LN will be asked to participate in this project, and will receive treatment according to current guidelines. Half of the patients will undergo a repeat biopsy 12 months later, and half of the patients will not. The selection of patients who will undergo or not undergo repeat biopsy will be random. Patients with high disease activity at the level of kidney tissue will receive more intense immunosuppressive treatment. Patients who have not undergone repeat biopsy will continue to be treated according to standard routine.

The investigators will compare the results of treatment between the group of patients who underwent and the group of patients who did not undergo repeat biopsy, with regard to (i) complete disease inactivity at month 24 and (ii) renal function at month 60 from treatment initiation.

The investigators expect that significantly greater proportions of patients in the repeat biopsy group will have inactive disease at month 24 and adequate levels of renal function at month 60. This will provide support for performing repeat biopsies as a part of the treatment evaluation, in order to optimise the therapeutic management and improve the long-term prognosis of patients with LN.

DETAILED DESCRIPTION:
Study rationale

Lupus nephritis (LN) affects 35-60% of patients with systemic lupus erythematosus (SLE), and constitutes one of the most severe disease manifestations. Several factors contribute to renal function impairment in LN, including genetic cargo, nephron endowment, disease activity, drug-induced toxicity and renal flares. Five to 20% of the afflicted patients develop end-stage kidney disease (ESKD) within ten years from the first LN episode. Available therapies induce complete renal remission in only 20-30% of patients after six months of treatment, and even patients who respond to therapy may relapse in 35% of the cases.

To date, clinical and laboratory tests cannot reliably reflect histopathological findings, and kidney biopsy is indispensable for diagnosis, classification, and exclusion of mimickers. The role of control biopsies after induction therapy is debatable, despite accumulating evidence of discrepancies between clinical and histological responses. In the concrete, several elegant post-treatment biopsy studies have demonstrated persistent activity at the level of tissue despite adequate clinical response, suggesting that intensified immunosuppression may be required in these patients. However, studies investigating the role of repeat kidney biopsies in treatment evaluation and long-term renal outcome have to date included limited numbers of patients, and varying definitions regarding treatment response and renal outcome. Thus, the concept of a prospective multicentric per-protocol repeat biopsy study to generate evidence for future recommendations for the diagnostic and therapeutic management of LN gains increasing support.

Several studies have sought to identify predictors of long-term renal prognosis, including routine clinical and serological markers. Proteinuria levels < 0.7-0.8 g/day at month 12 after initiation of treatment have been validated in different cohorts as a readily available predictor of favourable long-term renal outcome. However, while the positive predictive value (PPV) of this target was high, the negative predictive value (NPV) was poor in two of three studies, since most patients not achieving the proteinuria target still had a good long-term outcome (Tamirou et al. 2015; Ugolini-Lopes et al. 2017). Associations between chronic tissue damage in repeat biopsies and long-term renal function impairment have been demonstrated in European and Hispanic LN populations (Piñeiro et al. 2016). It was recently demonstrated in a retrospective study that a high grade of residual activity in per-protocol repeat biopsies predicted subsequent renal relapse in patients with incident LN, and a high grade of chronic damage in repeat biopsies predicted long-term renal function impairment. More specifically, NIH activity index scores > 3 predicted subsequent renal flares, whereas NIH chronicity index scores > 3 were associated with renal function deterioration in the long term. It is worth noting that active lesions in glomeruli mostly accounted for the former association with relapses, whereas chronic damage in the tubulointerstitial compartment were found to be a more important contributor to the latter association with long-term renal function (Parodis et al. 2020).

Study objectives

The objectives of the project will be

* to determine the percentage of LN patients in histopathological remission after 12 months of standard of care immunosuppression;
* to correlate histological and immunological (immune deposits) response to therapy with clinical response;
* to evaluate whether therapeutic decisions steered by the results of a per-protocol repeat kidney biopsy improve renal outcomes compared with a matched control group of patients who did not undergo repeat kidney biopsy.
* to generate data on how to evaluate response to therapy in pure membranous LN (ISN/RPS class V), as well as the value of the information retrieved from repeat kidney biopsies in portending long-term renal prognosis in this LN subset.

Study design

Patients with an incident biopsy-proven proliferative or membranous LN, or combinations thereof, selected to be initiated at standard of care immunosuppressive therapy with either MMF or EURO-Lupus IV CYC (combined with GCs and ACE inhibitors/ARBs) will be enrolled in this prospective study. Add-on therapies on the top of the aforementioned regimens will be allowed. At baseline, patients will be randomised 1:1 to either undergo or not undergo a per-protocol repeat kidney biopsy at month 12 from baseline. After randomisation, the patients will be followed for one year within the frame of REBIOLUP Part I, which is observational. Inclusion of patients participating in other investigator-initiated or pharmaceutical industry-driven therapeutic trials will be made possible, provided that those trials do not last more than 12 months. At month 12, REBIOLUP patients will enter into Part II, which is interventional and an interval of ± 1 month is allowed.

In patients with 2003 ISN/RPS class III/IV (± V) at baseline and an NIH activity index score > 3 (cut-off based on a recent proof-of-concept retrospective analysis) in the repeat kidney biopsy, the immunosuppressive therapy will be intensified based on the physician's and patient's shared decision (see recommendations below). In cases of pure membranous nephritis (ISN/RPS class V) at baseline which transformed to ISN/RPS class III/IV (± V) in the repeat biopsy, the same algorithm will be applied.

In patients with pure membranous (2003 ISN/RPS class V) LN in the repeat biopsy, individual assessment of the biopsy should steer the decision of treatment.

Patients who have not undergone a repeat biopsy will be treated according to standard clinical parameters. Percentages of complete renal response at month 24 and renal impairment at month 60 will be compared between the two study arms.

Patients randomised to the control arm (i.e. to not undergo per-protocol repeat biopsy) who underwent a repeat kidney biopsy upon clinical indication approximately at month 12 from baseline, e.g. due to primary non-response or worsening, will be analysed in the control arm (as per intention) for the primary analysis, and, additionally, together with the patients in the interventional arm in a secondary analysis.

Statistical power calculation and number of subjects needed

The anticipated frequency of CRR at month 24 in patients of the "no repeat biopsy" arm is 40%. The investigators consider that a difference of 20% in favour of the "repeat biopsy" arm would be clinically meaningful (i.e. a frequency of 60% CRR at month 24). To detect such a difference, with an α level of 0.05 and a power of 0.80, a number of 98 patients per arm is required. In order to take an anticipated 5% drop-out proportion into account, 206 patients with incident proliferative [2003 ISN/RPS class III/IV (A or A/C)] lupus nephritis will need to be enrolled. Patients with incident active membranous LN (2003 ISN/RPS class V) will also be enrolled in REBIOLUP; however, the target number of patients per arm will be based on proliferative cases only, since power calculation has been based on data from studies of proliferative LN.

Based on an anticipated yearly inclusion rate of 3-5 patients per year per centre, i.e. 6-10 patients during a 2-year period, approximately 20-30 centres of LN expertise will need to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the EULAR/ACR classification criteria of SLE.
* 18 years of age or above.
* Incident biopsy-proven proliferative or membranous LN, or combinations thereof (with UPCR ≥ 1 g/g), i.e. 2003 ISN/RPS class III (A or A/C) ± V, class IV (A or A/C) ± V, or class V.
* Consent to the possibility of a repeat kidney biopsy at month 12 from baseline.
* Initiation of the following treatment regimens:

  * intravenous pulses of methylprednisolone (total dose of 500-3000 mg);
  * oral prednisone or equivalent 0.3-0.5 mg/kg/day with tapering;
  * hydroxychloroquine unless contraindicated;
  * angiotensin-converting enzyme (ACE) inhibitors or angiotensin II receptor blockers (ARBs);
  * either one of mycophenolate mofetil (MMF) equivalent dose 2-3 g/day, or IV cyclophosphamide (CYC) according to the Euro-Lupus regimen;
  * the NIH protocol for IV CYC (0.5-0.75 g/m2 monthly for six months) could be considered in severe cases;
  * add-on therapies (e.g. calcineurin inhibitors, biologics) to the above two regimens are optional.

Exclusion Criteria:

* Antiphospholipid syndrome nephropathy (APSN).
* Pregnancy at baseline (pregnancy during follow-up will not lead to exclusion).
* Medical contraindications to kidney biopsy, e.g. thrombocytopenia < 50,000/μL, uncontrolled hypertension or end-stage kidney disease (ESKD).
* Anticipated non-adherence to therapy.
* Medical conditions interfering with outcome evaluations.
* Inability to read and/or sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Complete Renal Response (CRR) at month 24 from baseline | Month 24 from baseline
  UPCR ≤ 0.5 g/g in two consecutive first-morning void urine specimens and no increase in serum creatinine by ≥ 25% from baseline.

SECONDARY OUTCOMES:
Renal function impairment at month 60 | Month 60 from baseline
  Sustained (i.e. observed in at least two consecutive measurements on different dates) increase in serum creatinine by ≥ 25% from baseline.
Renal relapse (proteinuric flare) | Between month 12 and month 60 from baseline
  Reappearance of UPCR > 1.0 g/g from month 12 onwards, leading to intensification or change of immunosuppressive therapy. This increased proteinuria has to be sustained (i.e. observed in at least two consecutive measurements on different dates), occurring after an initial response to induction therapy (defined as sustained UPCR < 0.5 g/g).
Reabsorption of immune deposits in repeat kidney biopsies | Month 12 from baseline
  ≥ 50% decrease in intensity and amount of immune deposits in electron microscopy.
End-stage kidney disease (ESKD) | Between month 12 and month 60 from baseline
  Chronic kidney disease stage 5 and/or dialysis will be used to assess ESKD.
Mortality rate | Between month 12 and month 60 from baseline
  The number of deaths during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Parodis, MD PhD, Study Chair — Karolinska Institutet; Farah Tamirou, MD PhD, Study Chair — Université Catholique de Louvain; Julia Weinmann-Menke, MD PhD, Study Chair — Johannes Gutenberg University Mainz; Hans-Joachim Anders, Professor, Study Chair — Ludwig-Maximilians - University of Munich; Brad H Rovin, Professor, Study Chair — Ohio State University; Frédéric A Houssiau, Professor, Study Chair — Université Catholique de Louvain
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Datasets needed for addressing research questions that have not been addressed in the original publications.
Supporting Information: Study Protocol, ICF
Time Frame: Starting ten years after the baseline visit of the last study participant recruited.
Access Criteria: The REBIOLUP steering committee will review all proposals and provide IPD to investigators upon reasonable request, however highly depending on the research questions to be addressed.
URL: http://rebiolup.com

REFERENCES:
- [Background] Newman LB, Anderson EE, Waggover MD, Schulman CC. The relationship of blood urea nitrogen and serum uric acid: a computerized analysis. Acta Urol Belg. 1972 Oct;40(4):784-7. No abstract available. PMID 4654096
- [Background] Robertson DR. The ultimobranchila body in Rana pipiens. VII. Cellular responses in denervated glands in autoplastic transplants. Z Zellforsch Mikrosk Anat. 1968;90(2):273-88. No abstract available. PMID 5724342
- [Background] Pineiro GJ, Arrizabalaga P, Sole M, Abellana RM, Espinosa G, Cervera R. Repeated Renal Biopsy - A Predictive Tool to Assess the Probability of Renal Flare in Lupus Nephritis. Am J Nephrol. 2016;44(6):439-446. doi: 10.1159/000452229. Epub 2016 Oct 28. PMID 27788504
- [Background] Parodis I, Adamichou C, Aydin S, Gomez A, Demoulin N, Weinmann-Menke J, Houssiau FA, Tamirou F. Per-protocol repeat kidney biopsy portends relapse and long-term outcome in incident cases of proliferative lupus nephritis. Rheumatology (Oxford). 2020 Nov 1;59(11):3424-3434. doi: 10.1093/rheumatology/keaa129. PMID 32353879